CLINICAL TRIAL: NCT03434158
Title: Phase II Trial Evaluating Olaparib Maintenance in Patients With MCRPC After Docetaxel Treatment Reaching Partial or Stable Response.
Brief Title: Olaparib Maintenance in Patients With MCRPC After Docetaxel Treatment Reaching Partial or Stable Response (IMANOL)
Acronym: IMANOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: AstraZeneca (Industry); Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOGUG-2016-A-IEC(PRO)-12; 2017-001469-26 (EudraCT Number)
Record Dates: First submitted 2018-01-26; First posted 2018-02-15 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer Metastatic
Keywords: Metastatic Prostate Cancer Resistant to Castration
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olaparib (Experimental): 600 mg/day
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — 300 mg twice a day
  Other Names: Lynparza

SUMMARY:
A number of important systemic therapies have been developed to treat mCRPC and have received regulatory approval and now comprise the current therapeutic landscape. Durable and complete response following first-line chemotherapy in patients with advanced PC are uncommon. Most patients will ultimately experience disease progression within 6-9 months after initial response. Optimal Second line therapy in mCRPC is not well established and several options are possible.

Olaparib has demonstrated anti-tumour activity in non-comparative studies in patients with germline BReast CAncer gene (gBRCA) mutated cancers including ovarian, breast, pancreas and prostate. Olaparib is indicated as monotherapy for the maintenance treatment of adult patients with platinum-sensitive relapsed Breast Cancer gene-mutated (germline and/or somatic) high grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer who are in response (complete response or partial response) to platinum-based chemotherapy.

This phase II study is developed to assess the effect of maintenance treatment with olaparib on radiologic progression free survival (rPFS) in patients with mCRPC who have received at least 6 cycles of docetaxel and achieved partial or complete response or disease stabilization according RECIST 1.1 criteria and PCWG3.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures. For inclusion in the study patients must provide the informed consent also for genetic research. Genetic counselling for patients with germline mutation in any of the Homologous Recombination Repair genes should be performed.
* Male patients, who must be ≥18 years of age.
* Histologically confirmed prostate adenocarcinoma.
* Patients must have metastatic disease before starting treatment with docetaxel (metastatic disease documented by positive bone scan or metastatic lesions on CT, MRI).
* No prior exposure to platinum, cyclophosphamide, mitoxantrone or Polyadenosine 5'diphosphoribose polymerisation (PARP) inhibitors.
* No cancer progression on the basis of Prostate Cancer Working Group (PCWG3) criteria to docetaxel therapy.
* Completed at least six cycles and a maximum of ten cycles of chemotherapy containing docetaxel.
* Patients are allowed to have received treatment for mCRPC before docetaxel (abiraterone, enzalutamide, radium 223,etc.; patients that have received prior docetaxel in hormone-sensitive setting are also allowed).
* Documented germline/somatic mutation in any of the Homologous Recombination Repair genes, including among others, BRCA1 or BRCA2, ATM, Fanconi genes, CHEK2, mutL homolog 1 (MLH1), mutS homologue 2 (MSH2), mutS homolog 6 (MSH6), PMS2, PALB2, RAD51C, MRE11 that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function).
* Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

  * Haemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days.
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
  * Platelet count ≥ 100 x 109/L.
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
  * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase ((SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN.
  * Patients must have creatinine clearance estimated using the Cockcroft-Gault equation of ≥51 mL/min:

Estimated creatinine clearance = ((140-age [years]) x weight (kg) (x F)^a) / serum creatinine (mg/dL) x 72 F=1 for males.

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Patients must be able to take oral medication.
* Patients must have a life expectancy ≥ 16 weeks.
* Male patients and their partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination [see appendix A for acceptable methods], throughout the period of taking study treatment and for 3 months after last dose of study drug(s) to prevent pregnancy in a partner.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
* Formalin fixed, paraffin embedded (FFPE) tumour sample from the primary cancer must be available for central testing. If there is not written confirmation of the availability of an archived tumour sample prior to enrolment the patient is not eligible for the study.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to AstraZeneca or sponsor staff and/or staff at the study site).
* Previous inclusion in the present study.
* Participation in another clinical study with an investigational product during the last month.
* Any previous treatment with PARP inhibitor, including olaparib.
* Patients who do not have deleterious or suspected deleterious Homologous Recombination Repair genes mutations and only have Homologous Recombination Repair genes mutations that are considered to be non-detrimental (e.g., "Variants of uncertain clinical significance" or "Variant of unknown significance" or "Variant, favour polymorphism" or "benign polymorphism" etc.).
* Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma, or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years.
* Resting ECG with corrected QT interval (QTc) > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment.
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia and nail toxicity.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
* Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
* Major surgery within 4 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Patients with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids.
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Histologically confirmed prostate adenocarcinoma.
Enrollment: 16 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Radiographic progression free survival (rPFS) | Up to 1 year
  Time from treatment with olaparib to the date of first disease radiographic progression or death for any reason. Radiographic progression disease will be evaluated according RECIST 1.1 criteria and PCWG3

SECONDARY OUTCOMES:
PSA progression free survival (PSA PFS) | Up to 1 year
  Time from treatment with olaparib to the date of first PSA progression (according PWCG3 criteria) or death for any reason.
Clinical PFS | Up to 1 year
  Time from treatment with olaparib to the date of first clinical progression (significant pain increase or clinical deterioration that requires initiating another line of treatment) or death for any reason.
Radiologic response rate | Up to 1 year
  Radiographic response will be evaluated according RECIST 1.1.
PSA response rate | Up to 1 year
  PSA response is a reduction in serum PSA concentration of ≥50% from baseline.
Number of individual events (hematologic events and not hematologic events) | Up to 1 year
  Number of events per patient

OTHER OUTCOMES:
Gene mutation(s) | At Baseline
  Number of gene mutation/s

CONTACTS AND LOCATIONS:
Overall Officials: María J Juan Fita, MD, Principal Investigator — Fundación Instituto Valenciano de Oncología
Locations (8):
- Spain (8):
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clínic de Barcelona, Barcelona
  - Complejo Hospitalario Regional Reina Sofía, Córdoba
  - Hospital Universitario 12 de Octubre, Madrid
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Universitario i Politècnic La Fe, Valencia